CLINICAL TRIAL: NCT06621082
Title: A Prospective, One-arm, Phase II Clinical Study of Smeitinib Hydrosulfate Capsules for the Treatment of Patients With Type I Neurofibromatosis After Surgery
Brief Title: The Clinical Study of the Treatment of Patients With Type I Neurofibromatosis With Smetinib Hydrosulfate Capsule
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-284-02
Record Dates: First submitted 2024-08-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Postoperative drug group (Experimental): This study started from the recruitment of subjects, confirmed diagnosis by clinical diagnosis and pathological biopsy, preliminary screening according to inclusion and exclusion criteria, and signing of informed consent. Patients who were evaluated as indications for surgical resection and underwent surgical treatment were treated with Smetinib bisulfate capsules. PFS, ORR, and DOR were evaluated after 6 cycles of administration of Simetinib bisulfate capsules (20-50mg bid) daily for 30 days, as individualized by patient body surface area (BSA).
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — After surgical resection，based on the patient's body surface area (BSA), the patient was given an oral dose of Simetinib bisulfate capsule (20-50mg bid) daily for 30 days for 6 cycles

SUMMARY:
This study focused on patients with type I neurofibromatosis undergoing surgical treatment, who currently lack effective drug therapy and have a high recurrence rate after surgical resection. For patients with small solid tumors, limited space, and no invasion of the brain, spine and other important organs, surgical treatment is the main treatment. As a MEK inhibitor, Smetinib bisulfate capsule can induce tumor shrinkage and reduce postoperative recurrence by selectively binding mitogen-activated protein kinase (MEK) 1/2 protein to block the mitogen-activated protein kinase/extracellular signal regulatory kinase signaling pathway that regulates key cell responses. The purpose of this study was to treat patients with type I neurofibromatosis with indications of surgery with the drug smetinib bisulfate after surgical treatment, observe the therapeutic effect of the drug in stages, consolidate the postoperative effect and reduce the recurrence rate. In this study, progression-free survival (PFS) after postoperative drug treatment was used as the main outcome index, and duration of remission (DOR) and objective response rate (ORR) were used as secondary outcome indicators to investigate the efficacy of the use of Smetinib hydrosulfate capsule on tumor control, reduction of recurrence rate and stability of efficacy in patients with type I neurofibromatosis after surgery.

DETAILED DESCRIPTION:
Neurofibromatosis (NF) has been included in the list of rare diseases in many countries, including China, of which 96% is NF1 subtype, NF1 clinical manifestations are diverse, involve multiple systems, can cause respiratory obstruction, spinal cord compression, motor dysfunction and other serious complications. Plexiform neurofibroma (PN) occurs in 30-50% of patients with NF1. PN progresses rapidly, is associated with severe physical defects, is highly disabling, and is at risk of malignancy. According to the 2023 edition of the Multidisciplinary Guidelines for the Diagnosis and Treatment of type I neurofibromatosis, NF1 patients are more likely than the normal population to develop a variety of benign and malignant tumors, including pNF, CNF, MPNST and OPG. Attention should be paid to the early identification and monitoring of these tumors. The possibility of MPNST should be highly vigilant for neurofibromas with growth acceleration, pain, and texture hardening. At the same time, systemic evaluation should be performed, and early surgery should be performed as far as possible for patients without signs of distant metastasis, while radiotherapy, chemotherapy and targeted therapy can be selected for patients with distant metastasis.

neurofibromatosis type 1 (NF1) is an autosomal dominant disorder in which 50% of patients have familial inherited mutations and 50% have sporadic mutations. NF1 gene encodes neurofibrin, down-regulates the activity of Ras-Raf pathway, and inhibits cell proliferation. Neurofibrin defects can lead to overactivation of the RAS pathway, resulting in uncontrolled cell proliferation in patients with NF1. At present, surgery is the most commonly used and most important treatment for neurofibromatosis, and neurofibroma has the characteristic of growing along the nerve root, so it is difficult to solve all the lesions through surgery. The lesions consist of a wide range of nerve and vascular tissues mixed with normal tissues, and the surgical resection is difficult and bleeding is frequent, and the recurrence after incomplete resection is as high as 50%. For NF1 in the head and neck, some patients require a second operation one year after surgery, and the proportion of patients with partial resection undergoing a second operation is higher than that of patients with subtotal resection. Five years after surgery, more than 50% of patients needed a second operation.

As a MEK inhibitor, Smetinib bisulfate capsule can induce tumor shrinkage by selectively binding mitogen-activated protein kinase (MEK) 1/2 protein to block the mitogen-activated protein kinase/extracellular signal regulatory kinase signaling pathway that regulates key cellular responses. To create conditions for disease control, radical surgical resection, reducing postoperative recurrence and reducing complications. Based on the targeted therapy of smeitinib bisulfate capsule, this study evaluated the treatment of NF1 patients after surgical treatment, and evaluated the effect of tumor shrinkage after medication by monitoring the effect and duration of solid tumor shrinkage of patients. And the postoperative recurrence time, so as to verify the effectiveness of smeitinib bisulfate capsule in reducing the recurrence rate of patients after NF1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. According to the National Institutes of Health (NIH) updated diagnostic criteria for NF1 in 2021, 6 or more CALMs: d>5 mm before puberty or d>15 mm after puberty; 2 or more neurofibromas of any type or 1 plexiform neurofibroma;

   ③ Freckles in the armpit or groin area;

   ④ optic glioma (OPG);

   ⑤ Two or more Lisch nodules were detected by slit-lamp, or two or more choroidal abnormalities were detected by optical coherence tomography (OCT)/ near-infrared (NIR) imaging;

   ⑥ Characteristic bone lesions, such as sphenoid dysplasia, anterolateral tibial curvature; Pathogenic heterozygote NF1 variant with 50% allele variant fraction in normal tissues (such as white blood cells); NF1 is diagnosed in persons who have no history of parental disease and meet 2 or more clinical characteristics Individuals with a history of parental disease who meet one or more clinical characteristics may be diagnosed with NF1
3. Before admission, the head and neck surgeon conducted pathological biopsy of solid tumors, confirmed pathological diagnosis and eliminated malignant peripheral schwannoma (MPNST).
4. There was at least one measurable tumor lesion according to the solid tumor efficacy evaluation criteria RECIST 1.1
5. The tumor did not invade the brain, spine and other important organs, there are indications of surgical resection and surgical treatment
6. The performance of the Eastern Cooperative Oncology Group (ECOG) was 0-1
7. Blood routine: white blood cell count (WBC) ≥3.0×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet (PLT) ≥ 100×109/L; Hemoglobin level (HGB) ≥ 9.0 g/dL (7 days without corresponding supportive treatment, such as blood transfusion and increased white blood cells).
8. Liver function: the patient's aspartate aminotransferase (AST) and alanine aminotransferase (ALT) were less than 2.5 times the upper limit of reference value (ULN); Albumin (ALB) ≥ 30 g/L.
9. Renal function: serum creatinine ≤1.5 times ULN or creatinine clearance (CrCl) ≥ 50mL/min (using Cockcroft/Gault formula); Urinary protein (UPRO) < (++), or 24-hour urinary protein volume < 1.0 g.
10. Cardiac function: creatine phosphokinase ≤200U/L, left ventricular ejection fraction (LVEF) ≥50%;
11. Have not participated in other clinical trials within the past 30 days;
12. Patients who voluntarily participate in the project and sign informed consent.

Exclusion Criteria:

1. The patient had abnormal blood indexes and abnormal liver, kidney and heart function, and could not tolerate the clinical study process after multidisciplinary consultation and evaluation
2. The patient has become malignant peripheral schwannoma (MPNST) or is accompanied by other malignant tumors, heart disease and other serious complications, or has previously received chemotherapy, radiotherapy and other anti-tumor therapy
3. Unable to complete the entire clinical study due to personal, social and economic reasons
4. there is a serious systemic disease in the past and the disease cannot be cured or controlled by medicine at present
5. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival (2-year PFS rate) | Within 2 years from the start of treatment in the trial
  Refers to the rate of postoperative patients who are free of tumor progression or death from any cause (whichever occurs first) within 2 years from the start of treatment in the trial.

SECONDARY OUTCOMES:
Duration of remission | Within 2 years from the start of treatment in the trial
  Refers to the time from the first evaluation of a tumor as CR or PR to the first evaluation as PD or death from any cause
Objective response rate | Within 2 years from the start of treatment in the trial
  The proportion of patients whose tumors shrink by ≥ 20% for a certain period of time, including complete response (CR) and partial response (PR) cases. ORR was defined as the proportion of patients whose tumor size decreased by ≥ 20% in the shortest time.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiquan Huang, doctoral, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ly KI, Blakeley JO. The Diagnosis and Management of Neurofibromatosis Type 1. Med Clin North Am. 2019 Nov;103(6):1035-1054. doi: 10.1016/j.mcna.2019.07.004. PMID 31582003
- [Result] Gutmann DH, Ferner RE, Listernick RH, Korf BR, Wolters PL, Johnson KJ. Neurofibromatosis type 1. Nat Rev Dis Primers. 2017 Feb 23;3:17004. doi: 10.1038/nrdp.2017.4. PMID 28230061
- [Result] Di Rocc C, Samii A, Tamburrini G, Massimi L, Giordano M. Sphenoid dysplasia in neurofibromatosis type 1: a new technique for repair. Childs Nerv Syst. 2017 Jun;33(6):983-986. doi: 10.1007/s00381-017-3408-z. Epub 2017 Apr 13. PMID 28409229
- [Result] Miller DT, Freedenberg D, Schorry E, Ullrich NJ, Viskochil D, Korf BR; COUNCIL ON GENETICS; AMERICAN COLLEGE OF MEDICAL GENETICS AND GENOMICS. Health Supervision for Children With Neurofibromatosis Type 1. Pediatrics. 2019 May;143(5):e20190660. doi: 10.1542/peds.2019-0660. PMID 31010905
- [Result] Blakeley JO, Plotkin SR. Therapeutic advances for the tumors associated with neurofibromatosis type 1, type 2, and schwannomatosis. Neuro Oncol. 2016 May;18(5):624-38. doi: 10.1093/neuonc/nov200. Epub 2016 Feb 6. PMID 26851632
- [Result] Friedrich RE, Schmelzle R, Hartmann M, Funsterer C, Mautner VF. Resection of small plexiform neurofibromas in neurofibromatosis type 1 children. World J Surg Oncol. 2005 Jan 31;3(1):6. doi: 10.1186/1477-7819-3-6. PMID 15683544
- [Result] Prada CE, Rangwala FA, Martin LJ, Lovell AM, Saal HM, Schorry EK, Hopkin RJ. Pediatric plexiform neurofibromas: impact on morbidity and mortality in neurofibromatosis type 1. J Pediatr. 2012 Mar;160(3):461-7. doi: 10.1016/j.jpeds.2011.08.051. Epub 2011 Oct 11. PMID 21996156
- [Result] Martin S, Wolters P, Baldwin A, Gillespie A, Dombi E, Walker K, Widemann B. Social-emotional functioning of children and adolescents with neurofibromatosis type 1 and plexiform neurofibromas: relationships with cognitive, disease, and environmental variables. J Pediatr Psychol. 2012 Aug;37(7):713-24. doi: 10.1093/jpepsy/jsr124. Epub 2012 Feb 21. PMID 22353803
- [Result] Ferner RE, Huson SM, Thomas N, Moss C, Willshaw H, Evans DG, Upadhyaya M, Towers R, Gleeson M, Steiger C, Kirby A. Guidelines for the diagnosis and management of individuals with neurofibromatosis 1. J Med Genet. 2007 Feb;44(2):81-8. doi: 10.1136/jmg.2006.045906. Epub 2006 Nov 14. PMID 17105749
- [Result] Anderson MK, Johnson M, Thornburg L, Halford Z. A Review of Selumetinib in the Treatment of Neurofibromatosis Type 1-Related Plexiform Neurofibromas. Ann Pharmacother. 2022 Jun;56(6):716-726. doi: 10.1177/10600280211046298. Epub 2021 Sep 18. PMID 34541874
- [Result] Harder A. MEK inhibitors - novel targeted therapies of neurofibromatosis associated benign and malignant lesions. Biomark Res. 2021 Apr 16;9(1):26. doi: 10.1186/s40364-021-00281-0. PMID 33863389
- [Result] Campagne O, Yeo KK, Fangusaro J, Stewart CF. Clinical Pharmacokinetics and Pharmacodynamics of Selumetinib. Clin Pharmacokinet. 2021 Mar;60(3):283-303. doi: 10.1007/s40262-020-00967-y. Epub 2020 Dec 23. PMID 33354735
- [Result] Gross AM, Wolters PL, Dombi E, Baldwin A, Whitcomb P, Fisher MJ, Weiss B, Kim A, Bornhorst M, Shah AC, Martin S, Roderick MC, Pichard DC, Carbonell A, Paul SM, Therrien J, Kapustina O, Heisey K, Clapp DW, Zhang C, Peer CJ, Figg WD, Smith M, Glod J, Blakeley JO, Steinberg SM, Venzon DJ, Doyle LA, Widemann BC. Selumetinib in Children with Inoperable Plexiform Neurofibromas. N Engl J Med. 2020 Apr 9;382(15):1430-1442. doi: 10.1056/NEJMoa1912735. Epub 2020 Mar 18. PMID 32187457
- [Result] Dombi E, Baldwin A, Marcus LJ, Fisher MJ, Weiss B, Kim A, Whitcomb P, Martin S, Aschbacher-Smith LE, Rizvi TA, Wu J, Ershler R, Wolters P, Therrien J, Glod J, Belasco JB, Schorry E, Brofferio A, Starosta AJ, Gillespie A, Doyle AL, Ratner N, Widemann BC. Activity of Selumetinib in Neurofibromatosis Type 1-Related Plexiform Neurofibromas. N Engl J Med. 2016 Dec 29;375(26):2550-2560. doi: 10.1056/NEJMoa1605943. PMID 28029918

DOCUMENTS (1):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT06621082/Prot_000.pdf